CLINICAL TRIAL: NCT01067196
Title: A Study of Late Effects After Proton Radiotherapy for Pediatric Tumors of the Brain, Head, and Neck
Brief Title: Outcomes Study of Late Effects After Proton RT for Pediatric Tumors of the Brain, Head, and Neck
Acronym: CN01
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201701741; UFPTI 0903-CN01 (Other: University of Florida Project #)
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Central Nervous System Tumors
Keywords: Proton Radiation; Central Nervous System (CNS) Tumors; Brain; Spine; Cancer; Radiation Therapy (RT)
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation and quality of life: Central Nervous System Tumors

SUMMARY:
The purpose of this study is to collect information from medical records to see what effects proton beam radiation has on cancer and analyze possible side effects.

DETAILED DESCRIPTION:
Data collection will be obtained from the patient's medical records including initial evaluation, radiotherapy completion records and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Estimated >5 cc of the brain tissue to receive >5 CGE radiation
* Patient must be less than 21 years of age at time of consent.
* Patients that require localized and craniospinal irradiation.
* Patients and/or patient parent must complete baseline Quality of Life Questionnaire as applicable by patient age group.

Exclusion Criteria:

* Prior radiation therapy.
* Evidence of metastases outside the central nervous system.

Ages: 1 Day to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients treated at a radiation oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Measure late effects of proton therapy on pediatric patients with CNS tumors | 5.4 years after treatment completion

SECONDARY OUTCOMES:
Survival endpoints of local control, progression-free survival, and overall and cause-specific survival. | 12 years after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Indelicato, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

REFERENCES:
- [Background] Duffner PK, Horowitz ME, Krischer JP, Friedman HS, Burger PC, Cohen ME, Sanford RA, Mulhern RK, James HE, Freeman CR, et al. Postoperative chemotherapy and delayed radiation in children less than three years of age with malignant brain tumors. N Engl J Med. 1993 Jun 17;328(24):1725-31. doi: 10.1056/NEJM199306173282401. PMID 8388548
- [Background] Sklar CA, Constine LS. Chronic neuroendocrinological sequelae of radiation therapy. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1113-21. doi: 10.1016/0360-3016(94)00427-M. PMID 7713777
- [Background] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Background] Bhat SR, Goodwin TL, Burwinkle TM, Lansdale MF, Dahl GV, Huhn SL, Gibbs IC, Donaldson SS, Rosenblum RK, Varni JW, Fisher PG. Profile of daily life in children with brain tumors: an assessment of health-related quality of life. J Clin Oncol. 2005 Aug 20;23(24):5493-500. doi: 10.1200/JCO.2005.10.190. PMID 16110009
- [Background] Huang E, Teh BS, Strother DR, Davis QG, Chiu JK, Lu HH, Carpenter LS, Mai WY, Chintagumpala MM, South M, Grant WH 3rd, Butler EB, Woo SY. Intensity-modulated radiation therapy for pediatric medulloblastoma: early report on the reduction of ototoxicity. Int J Radiat Oncol Biol Phys. 2002 Mar 1;52(3):599-605. doi: 10.1016/s0360-3016(01)02641-4. PMID 11849779